CLINICAL TRIAL: NCT05742893
Title: Comparison of a Speech-Language Pathology Assessment Tool for Pragmatic and Discourse Skills for Patients With Schizophrenic Spectrum Disorders and Other Psychotic Disorders
Brief Title: Comparison of a Speech-Language Assessment Tool for Pragmatic and Discourse Skills in Schizophrenia Spectrum Disorders
Acronym: VEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-AOI-04
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic (Experimental): all patients have the study test
  Interventions: Diagnostic Test: Measurement of pragmatic and discourse test scores in the two scales.

INTERVENTIONS:
Diagnostic Test: Measurement of pragmatic and discourse test scores in the two scales. — The aim of this study is to compare the effectiveness of a newly developed speech-language assessment tool for pragmatic and discourse skills for patients suffering from schizophrenia .

SUMMARY:
The scientific literature has largely objectified language disorders in schizophrenia. And more precisely, the impairment of pragmatic and discursive language skills. Currently, there is no standardized language assessment tool specific to these patients. The aim of this study is to compare the effectiveness of a newly developed speech-language assessment tool for pragmatic and discourse skills for patients suffering from schizophrenia .

DETAILED DESCRIPTION:
The scientific literature has largely objectified language disorders in schizophrenia. And more precisely, the impairment of pragmatic and discursive language skills. Currently, there is no standardized language assessment tool specific to these patients. The aim of this study is to compare the effectiveness of a newly developed speech-language assessment tool for pragmatic and discourse skills for patients suffering from schizophrenia.

To do so, patients will have to pass six tests: three tests of the new tool and three corresponding gold standard tests. The first two tests will assess pragmatic skills by means of a semi-directed interview. The next two tests will assess discourse skills through two image description tasks. Finally, the last two tests will evaluate narrative skills through the oral restitution of two heard texts.

The main objective is to compare the performance of schizophrenic patients detected in the pathological zone with the scales of the new tool versus the gold standard scales.

The secondary objective is to determine which skills are most affected by comparing patients' scores in pragmatic skills versus those in discourse skills.

This tool would allow to precisely objectify language disorders and to optimize the multidisciplinary diagnosis and care of patients suffering from schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 60
* Patient with a diagnosis of schizophrenic spectrum disorder and other psychotic disorders meeting DSM V criteria
* Patient who has been clinically and treatment stable for at least three months
* Patient who can read and write French
* Patient who is a beneficiary of a social security plan or similar
* Patient with ability to sign free and informed consent

Exclusion Criteria:

* - Patient hospitalized under restraint
* Patient under guardianship
* Patient who has stopped taking his or her treatment
* Patient who had a change in treatment in the period of less than three months prior to the pass
* Patient with a worsening of the disease in the three months prior to the inclusion visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
assess of pragmatic skills | day 0
  The patients is evaluated by means of a semi-directed interview
assess discourse skills | day 0
  he patient is evaluated through two image description tasks
assess narrative skills | day 0
  the patients is evaluated through the oral restitution of two heard texts.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Michel, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No